CLINICAL TRIAL: NCT03222544
Title: Efficacy and Safety of Methylene Blue -Mediated Photodynamic Therapy for Diabetic Lower Limb Ulcer : a Randomized Controlled Study
Brief Title: Clinical Study of Methylene Blue - Mediated Photodynamic Therapy for Diabetic Lower Limb Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Cheng Qing-feng, Associate professor, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDT2017
Record Dates: First submitted 2017-07-05; First posted 2017-07-19 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Extremity Lower Ulcers
Keywords: methylene blue; Photodynamics Therapy
MeSH Terms: interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photodynamic Therapy (Experimental): The photosensitizer, methylene blue, is applied topically to the ulcer surface and the ulcer was shielded from light for 15 min. Then the ulcer area is illuminated using a photon therapy instrument for 20 minutes. Photodynamic therapy is applied once a day for a total of seven times.
  Interventions: Combination Product: methylene blue
- Photon therapy (Active Comparator): The placebo is applied topically to the ulcer surface and the ulcer was shielded from light for 15 min. Then the ulcer area is illuminated using a photon therapy instrument for 20 minutes. Photon therapy is applied once a day for a total of seven times.
  Interventions: Combination Product: Photon therapy instrument

INTERVENTIONS:
Combination Product: methylene blue — Continue treatment after 5mins suspension if the patient feels that the local temperature is too high to stand
  Arms: Photodynamic Therapy
Combination Product: Photon therapy instrument — Continue treatment after 5mins suspension if the patient feels that the local temperature is too high to stand
  Arms: Photon therapy

SUMMARY:
The investigators designed this prospective, randomized control study to confirm the efficacy and safety of methylene blue - mediated photodynamic therapy for diabetic lower limb ulcer and to explore its mechanism.

DETAILED DESCRIPTION:
OBJECTIVE- Infection is associated with poor healing of diabetic lower limb ulcer. Diabetic lower limb ulcer are often lower extremity vascular stenosis or occlusion, poor blood supply, making local ulcer local antibacterial drugs difficult to effectively reach and distribution, resulting in systemic antibacterial efficacy is limited, and easy to induce bacterial resistance at the same time . In recent years, the incidence of clinical multidrug-resistant bacteria increased, increasing the difficulty and cost of treatment.

The current study attempts to identify whether the photodynamic therapy (PDT) would kill the surface of ulcer bacteria and promote ulcer healing, and explore the mechanism of methylene blue-mediated photodynamic therapy for diabetic lower limb ulcer RESEARCH DESIGN AND METHODS-This study evaluated six clinical indicators： diabetic foot ulcer area reduction rate, inflammation control rate, Local bacterial load, the dose and use time of antibiotics, adverse reaction rate, bacterial biofilm,local neutrophil extracellular traps. The efficacy and safety of PDT could be confirmed if the clinical indicators of PDT group is better than the control group. In this study, three methods were used to investigate the mechanism of -methylene blue mediated photodynamic therapy for diabetic lower limb ulcer: a comparison of the bacterial load, bacterial biofilm,local neutrophil extracellular traps of the ulcer immediately pre-treatment and immediately,1-week ,2 week,1 momth post-treatment ; EXPECTED RESULTS-The investigators will expect that methylene blue-mediated photodynamic therapy could kill bacteria on the surface of diabetic lower limb ulcer and accelerate wound healing.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understand the whole test process, voluntary and signed informed consent form.
* 2. Men and women aged 18 to 80 years old.
* 3. Diagnosed with diabetic lower limb ulcer.
* 4. Ulcer duration> 1 month of wagner grade Ⅱ, Ⅲ subjects.
* 5. An ulcer area ≤100 cm² or of linear dimension ≤ 10 cm.

Exclusion Criteria:

* 1. Diagnosis of systemic infection or any concomitant infection that would require treatment with an additional antimicrobial agent.
* 2. Pregnant or lactating women.
* 3. Wagner grade Ⅰ, Ⅳ, Ⅴ subjects.
* 4. Patients with a peripheral vascular disease require immediate revascularization, and/or an ankle brachial systolic blood pressure (SBP) index<0.5 in the infected limb.
* 5. Patients with inappropriate health to participate as determined by the principal investigators.
* 6. Patients in the hepatitis A, hepatitis B, AIDS, tuberculosis and other infectious diseases of the active period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-29 (Estimated); Primary Completion 2020-04-29 (Estimated); Study Completion 2020-06-29 (Estimated)

PRIMARY OUTCOMES:
Change from baseline （Ulcer area）in the diabetic lower limb ulcer at day 7 | Baseline and day 7
  Changes of ulcer area before and after treatment
Change from baseline (immediately before the first treatment) in the bacterial load of the ulcer at one hour (immediately after the first treatment) | Baseline and (immediately after the first treatment)，day 7,14,21,28
  Changes of local bacterial load before and after treatment
Change from baseline(bacterial biofilm） | Baseline and day 7,14,21,28
  Changes of local bacterial biofilm before and after treatment

SECONDARY OUTCOMES:
The dose of antibiotics | 7 days during treatment
  Dosage of antibiotics during treatment
The time of antibiotics | 7 days during treatment
  Antibiotic use time during treatment
Adverse events | 7 days during treatment
  including pain,redness, and swelling
A comparison of local NET neutrophil extracellular traps before the first treatment and after the tenth treatment | Baseline and day 7,14,21,28
  Fluorescence intensity and area of local NET
Inflammation control rate | 7 days during treatment
  Duration of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Cheng, PhD, Principal Investigator — the First Affiliated Hospital, Chongqing Medical University, China
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tardivo JP, Adami F, Correa JA, Pinhal MA, Baptista MS. A clinical trial testing the efficacy of PDT in preventing amputation in diabetic patients. Photodiagnosis Photodyn Ther. 2014 Sep;11(3):342-50. doi: 10.1016/j.pdpdt.2014.04.007. Epub 2014 May 9. PMID 24814697
- [Result] Lei X, Liu B, Huang Z, Wu J. A clinical study of photodynamic therapy for chronic skin ulcers in lower limbs infected with Pseudomonas aeruginosa. Arch Dermatol Res. 2015 Jan;307(1):49-55. doi: 10.1007/s00403-014-1520-4. Epub 2014 Nov 20. PMID 25410983
- [Result] Detty MR, Gibson SL, Wagner SJ. Current clinical and preclinical photosensitizers for use in photodynamic therapy. J Med Chem. 2004 Jul 29;47(16):3897-915. doi: 10.1021/jm040074b. No abstract available. PMID 15267226
- [Result] Giraudeau C, Moussaron A, Stallivieri A, Mordon S, Frochot C. Indocyanine green: photosensitizer or chromophore? Still a debate. Curr Med Chem. 2014;21(16):1871-97. doi: 10.2174/0929867321666131218095802. PMID 24350844
- [Result] Nicolau DP, Stein GE. Therapeutic options for diabetic foot infections: a review with an emphasis on tissue penetration characteristics. J Am Podiatr Med Assoc. 2010 Jan-Feb;100(1):52-63. doi: 10.7547/1000052. PMID 20093545